CLINICAL TRIAL: NCT00282581
Title: A Phase 1, Double-Blind, Placebo-Controlled Study to Assess the Safety and Immunogenicity of MVA3000 Modified Vaccinia Ankara (MVA) Smallpox Vaccine in Vaccinia-Naive Human Immunodeficiency Virus (HIV)-Seropositive Subjects
Brief Title: Safety Study of MVA Smallpox Vaccine in HIV-positive Subjects Who Are Vaccinia Naive
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Senior managemnt decision
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: H-249-004
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections; Smallpox
Keywords: HIV; Smallpox; MVA
MeSH Terms: conditions — HIV Infections; Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- placebo (Placebo Comparator)
  Interventions: Biological: MVA Smallpox Vaccine

INTERVENTIONS:
Biological: MVA Smallpox Vaccine — 0.5mL of MVA3000 Smallpox Vaccine, 2 doses, separated by 28 days.
  Other Names: placebo

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of two MVA smallpox vaccine injections in healthy adults that are 18-35 years of age with HIV infection

DETAILED DESCRIPTION:
This is a multi-center study 90 HIV-seropositive subjects. There will be an injection of MVA smallpox vaccine or placebo on day 0 and day 28.

Subjects will be enrolled and vaccinated in two cohorts according to CD4 cell count levels and number of subjects vaccinated. Excluding the screening period, the study duration will be approximately 56 days with a follow up safety visit at study day 148 and a telephone health status interview at study day 208.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old and who were born after 1971 who have never had a smallpox vaccination or exposure to a vaccinia-containing product
* Subjects must test positive for HIV infection
* Subjects must be in good general health except for HIV infection, including no AIDS-defining illnesses.
* Female Subjects must not be pregnant or lactating, and all subjects must agree to practice birth control
* subjects must be clinically stable for 6 months prior to study enrollment.

Exclusion Criteria:

* Subjects with a known or suspected history of immunodeficiency (with the exception of HIV infection)
* Subjects with history or prior exposure to a vaccinia-containing product
* subjects with current radiation treatment or use of immunosuppressive or antineoplastic drugs (with exceptions)
* Subjects with concomitant illnesses associated with impairment of immunologic function.
* subjects with dementia
* Subjects with malignancy.
* Subjects with a known history of Cardiac disease, or who have risk factors for ischemic coronary disease, or other abnormalities
* Current or past history of eczema
* known allergies to any component of MVA, including eggs or egg products, or allergies to blood products
* females must not be pregnant and using approved contraceptives.
* Morbid obesity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety | Study Completion

SECONDARY OUTCOMES:
Immunogenicity | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Fischl, MD, Principal Investigator — University of Miami AIDS clinical research unit; Rafael E Campo, MD, Principal Investigator — University of Miami; Cecilia Shikuma, MD, Principal Investigator — University of Hawaii- Honolulu; Daniel Pearce, DO, Principal Investigator — AltaMed Health Services, Los Angeles; Jacob Lalezari, MD, Principal Investigator — Quest Clinical Research, San Francisco; Scott D Parker, MD, Principal Investigator — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AltaMed Health Services Corporation, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - University of Miami AIDS Clinical Research Unit, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of Hawaii, Honolulu, Hawaii

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com